CLINICAL TRIAL: NCT05240079
Title: Evaluation of Concordance Between the Measurements Obtained by an Acquisition System of Physiological Parameters (Heart Rate/SpO2) Via a Teleconsultation Camera System With Reference to Standard Acquisition Measurements
Brief Title: Evaluation of a New System for Heart Rate and SpO2 Measurement.
Acronym: CARDIASENS_2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A02217-34
Record Dates: First submitted 2022-01-19; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2021-11

CONDITIONS: Telemedicine
Keywords: Telemedicine; Heart rate; photoplethysmography
MeSH Terms: interventions — Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Device: Heart rate measurement with Caducy system (twice). SpO2 measurement with Caducy system (Twice).

INTERVENTIONS:
Device: Heart rate measurement with Caducy system (twice). SpO2 measurement with Caducy system (Twice). — Heart rate and SpO2 measurement with Caducy (the visage of the subject is filmed 30 seconds and 1 minute with a camera) and heart rate and SpO2 measurement with gold standard (heart rate monitor and oximeter pod linked to an acquisition station). The procedure is repeated twice.
  Other Names: Heart rate measurement with gold standard system (twice). SpO2 measurement with gold standard system (twice).

SUMMARY:
Caducy is a new medical device that is able to estimate physiological number such as heart rate and SpO2 via laptop or computer camera. The goal of this study is to evaluate the concordance of Caducy system in reference to gold standard which is a heart rate monitor and an oximeter pod linked to a station of acquisition regardless the human variability. The Caducy system measurement via camera is made by filming the visage of the patient during 1 minute.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or over.
* Patient affiliated to a social security scheme.
* Having received complete information on the organization of the research.
* Able to understand the requirements of the trial and having signed a free and informed consent prior to entering the study
* Patient taken care of by the CUMSAPA (Centre Universitaire de Médecine du Sport et Activité Physique Adaptées) service for an PFT (pulmonary function test), stress test, consultation of adapted physical activity or other functional explorations carried out by the service.
* Patient having carried out a preliminary clinical examination.

Exclusion Criteria:

* Acute phenomenon contra-indicating the performance of an PFT, stress test or other functional exploration.
* Person with tremors at the time of clinical examination (Parkinson, spasms...)
* People who cannot present the palms of both hands (amputation).
* Woman of childbearing age who does not have effective contraception.
* Person referred to in Articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code: Pregnant woman, parturient or nursing mother, Minor (non-emancipated), Adult person subject to a legal protection measure (guardianship, curatorship, safeguard of justice), Person of full age unable to express consent
* Persons deprived of their liberty by a judicial or administrative decision, persons undergoing psychiatric treatment under Articles L. 3212-1 and L. 3213-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2023-09-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
Caducy's heart rate measurement compared to standard | through study completion, an average of 6 month
  Heart rate (bpm) taken with gold standart Heart rate (bpm) calculated by CADUCY

SECONDARY OUTCOMES:
Caducy's SpO2 measurement compared to standard | through study completion, an average of 6 month
  Blood oxygen saturation (%) taken by gold standard Blood oxygen saturation (%) calculated by CADUCY